CLINICAL TRIAL: NCT06622668
Title: Phase 1/2 Multicenter, Open-label Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NTLA-3001 in Participants with Alpha-1 Antitrypsin Deficiency (AATD)-Associated Lung Disease
Brief Title: NTLA-3001 in Adults with Alpha-1 Antitrypsin Deficiency-Associated Lung Disease
Acronym: AATD
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Clinical trial ITL-3001-CL-101 for the investigational product NTLA-3001 was withdrawn due to prioritization of other Sponsor programs.
Sponsor: Intellia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITL-3001-CL-101
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Lung Disease; Pulmonary Disease; AATD; Alpha-1 Antitrypsin Deficiency; Alpha-1 Antitrypsin Deficiency-associated Lung Disease
Keywords: AATD
MeSH Terms: conditions — Lung Diseases; alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: Biological NTLA-3001

INTERVENTIONS:
Biological: Biological NTLA-3001 — IV administration of AAV and CRISPR/Cas9 gene editing system

SUMMARY:
This study will be conducted to evaluate the safety, tolerability, clinical activity, pharmacokinetics, and pharmacodynamics of NTLA-3001 in adults with alpha-1 antitrypsin deficiency (AATD) -associated lung disease

DETAILED DESCRIPTION:
This study consists of 2 parts: Phase 1 is an open-label, single-arm ascending dose study to characterize the safety and activity of NTLA3001 and identify the dose for evaluation in Phase 2. Phase 2 will follow as an open-label, dose expansion study to further characterize the safety and clinical activity of NTLA-3001 and provide an initial assessment of the effect of NTLA-3001 on clinical measures of pulmonary function.

ELIGIBILITY:
Inclusion:

1. Age 18 years to 75 years
2. Diagnosis of AATD ZZ/ZNull genotypes
3. FEV1 ≥35% and ≤65%
4. No evidence of liver cirrhosis
5. Adequate chemistry and hematology measures at screening
6. Participants must agree not to participate in another interventional study for the duration of this trial.
7. Participants must be capable of providing signed informed consent

Exclusion Criteria:

1. AATD genotypes outside of ZZ or ZNull
2. Participants with total antibodies to adeno-associated virus (AAV) serotype above laboratory assay cut off
3. Participants who have known negative reaction or hypersensitivity to any lipid nanoparticles (LNP) component.
4. Any condition that, in the Investigator's opinion, could adversely affect the safety of the participant.
5. Unwilling to comply with study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-01-09 (Estimated); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | From NTLA-3001 infusion up to week156 post infusion
  To evaluate the safety and tolerability of NTLA-3001 as determined by adverse events (AEs) and dose limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Pharmacodynamics | From NTLA-3001 infusion up to week 156 post infusion
  To evaluate the PD effect of NTLA-3001
Immune Response | From NTLA-3001 infusion up to week 156 post infusion
  To evaluate the immune response to NTLA-3001
Vector Shedding | From NTLA-3001 infusion up to week 156 post infusion, only during phase 2.
  To evaluate vector shedding following administration of NTLA-3001

CONTACTS AND LOCATIONS:
Locations (1):
- New Zealand Clinical Research, Aukland, New Zealand

IPD SHARING:
Plan to Share IPD: No